CLINICAL TRIAL: NCT05033392
Title: An Open, Single-center, Phase II Clinical Trial Evaluating the Efficacy of PD-1 Antibody (JS001) in Combination With Neoadjuvant Chemotherapy for Gastric/Gastroesophageal Junction Cancer
Brief Title: PD-1 Blockade With JS001 Plus Neoadjuvant Chemotherapy for Gastric/Gastroesophageal Junction Cancer
Acronym: PNACGEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wan He (Other)
Responsible Party: Sponsor-Investigator, Wan He, Principal Investigator, Shenzhen People's Hospital
Organization: Shenzhen People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNACGEC
Record Dates: First submitted 2021-08-03; First posted 2021-09-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Stomach Neoplasms
Keywords: PD-1 antibody; neoadjuvant chemotherapy; gastric cancer; gastroesophageal junction cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab group (Experimental): Toripalimab is administrated with160mg and repeated every 2 weeks.
  Interventions: Drug: Toripalimab Injection

INTERVENTIONS:
Drug: Toripalimab Injection — A domestic PD-1 antibody
  Other Names: JS001

SUMMARY:
Gastric cancer (GC),including cardia and noncardia gastric cancer, is responsible for over 480,000 new cases in 2020 and an estimated 370,000 deaths, making it the third most frequently diagnosed cancer and the third leading cause of cancer death in China. Majority of patients(63%) are presented with locally advanced gastric cancer (stage Ⅱ/Ⅲ) and the prognosis is poor. Previous studies have shown that patients with pathological complete response(pCR) following neoadjuvant therapy have longer survival. In 2019, Lancet Oncology published the FLOT4-AIO study which testified that perioperative chemotherapy with FLOT (5-FU/LV, oxaliplatin and docetaxel) regimen has improved pCR rate and prolonged progression free survival(PFS) and overall survival(OS) in patients with stage II/III gastric cancer. Moreover, PD-1 blockade such as nivolumab or pembrolizumab in combination with chemotherapy has shown higher objective response rate(ORR) as compared to chemotherapy alone in advanced gastric cancer. The nanoparticle albumin-bound paclitaxel has been recommended as the second-line chemotherapy for unresectable or recurrent gastric cancer based on the Chinese Society of Clinical Oncology(CSCO) guideline. When PD-1 antibody is applied, albumin-bound paclitaxel is considered as a better partner since no pretreatment of corticosteroids is needed. Thus, the investigators plan to conduct a phase II clinical trial to evaluate the efficacy and safety of toripalimab (PD-1 antibody) combined with the FLOAP (albumin-bound paclitaxel, oxaliplatin, fluorouracil and leucovorin) regimen as the perioperative treatment of cT2-4 and/or N+ GC. The primary end point is pCR rate. The secondary end points include disease free survival(DFS), OS, ORR, R0 resection rate, incidence of adverse events(AE).

DETAILED DESCRIPTION:
This phase Ⅱ trial is a single-arm, open-label, non-randomized and single center clinical study. Patients who met the inclusion criteria will receive the combination of toripalimab (160mg, iv, d1,q2w) with FLOAP (fluorouracil,2600mg/m2; leucovorin, 200mg/m2; oxaliplatin, 85mg/m2; albumin paclitaxel, 150mg/m2, d1, q2w) up to four cycles. After the fourth cycle of the treatment, the clinical efficacy and operation feasibility will be evaluated by the MDT discussions. And then, surgery will be performed within 4 weeks. After the surgery, patients will receive 4-cycle treatments of toripalimab combined with FLOAP regimen. The primary end point is pCR rate. The secondary end points included DFS, OS, ORR, R0 resection rate, incidence of AE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 yeas and ≤79 years. The gender is not limited.
2. Confirmed gastric and gastroesophageal junction adenocarcinoma by Gastroscopic biopsy histopathological examination.
3. Endoscopic ultrasonography and/or enhanced CT/MRI examination confirmed at the stage of cT3/4a Nx or T2 N1-3, M0(AJCC 8th) before randomization.
4. At least 15 unstained sections of formalin-fixed paraffin-embedded tumor tissue sections or fresh tumor tissues can be provided for PD-L1, TMB, tumor infiltrating T lymphocytes, MSI-H/dMMR and EBV detection.
5. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1
6. Adequate bone marrow and organ function meets the following criteria:

   1. Neutrophil count (ANC)≥1.5×l09/L
   2. Platelet (PLT) ≥80×109/L
   3. Hemoglobin (Hb) level ≥9.0 g/L
   4. Total bilirubin level≤1.5×ULN
   5. Alanine aminotransferase (ALT) level≤3×ULN
   6. Aspartate aminotransferase (AST) level ≤3×ULN
   7. International normalized value (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN
   8. Serum creatinine (Cr) level ≤1.5×ULN
   9. Creatinine clearance >50 ml/min (Calculated according to the Cockcroft-Gault formula)

Exclusion Criteria:

1. Patients with a history of severe hypersensitivity to other monoclonal antibodies or any component of toripalimab injection (JS001).
2. Preoperative pathology diagnosed as squamous cell carcinoma or neuroendocrine tumor.
3. Patients have experienced or currently have other malignancies within 5 years.
4. Patients have received prior therapy with anti-PD-1, anti-PD-L1 or anti-CTLA4 agent.
5. Patients with history of autoimmune disease; patients with autoimmune-related hypothyroidism receive stable doses of thyroid hormone replacement therapy Eligible to participate in this study; Type 1 diabetes patients who are controlled after receiving a stable insulin treatment plan are eligible to participate in this study;
6. Patients have received systemic immunostimulatory drug therapy (including but not limited to interferon or IL-2) within 4 weeks before enrollment or within 5 half-lives of the drug (whichever is shorter);
7. Patients who have undergone allogeneic bone marrow transplantation or solid organ transplantation in the past;
8. Active infections, including tuberculosis (clinical diagnosis includes clinical history, physical examination and imaging findings, and TB examination according to local medical routines), hepatitis B {known HBV surface antigen (HBsAg) positive, and HBV DNA ≥1000cps/ml}, hepatitis C or human immunodeficiency virus (HIV antibody positive).
9. Patients with previous or cured HBV infection (defined as hepatitis B core antibody [anti-HBc] positive and HbsAg negative) are only eligible to participate in this study when HBV DNA is negative (HBV DNA ˂1000cps/ml).
10. Patients with positive hepatitis C (HCV) antibodies are only eligible to participate in this study if the polymerase chain reaction shows negative HCV RNA.
11. There is a serious neurological or mental illness, including dementia and seizures.
12. Suffer from NCI-CTCAE ≥ Grade 2 peripheral neuropathy.
13. Women who are pregnant or breastfeeding.
14. Chronic bowel disease or short bowel syndrome.
15. Those who are deficient in the enzyme dihydropyrimidine dehydrogenase (DPD).
16. Major cardiovascular diseases, such as New York Heart Association heart disease (level II or higher), myocardial infarction within 3 months before randomization, unstable arrhythmia, or unstable angina.
17. Patients with known coronary artery disease, congestive heart failure that does not meet the above criteria, or left ventricular ejection fraction <50% must adopt an optimized and stable medical plan determined by the treating doctor. If necessary, you can consult a cardiologist.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | Up to 6 months
  The proportion of patients with no tumor cells in the postoperative specimens

SECONDARY OUTCOMES:
Disease Free Survival | Up to 5 years
  Time from the date of treatment administration until the date of the first documented event of: disease recurrence following surgery (preferably biopsy proven), or death - whichever occurs first
Overall Survival | Up to 5 years
  Overall survival is defined as time from the date of treatment administration until the date of death from any cause.
Objective Response Rate | Up to 6 months
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
R0 Resection Rate | Up to 6 months
  Rate of microscopically margin-negative resection
Incidence of Adverse Events | Up to 6 months
  Number of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), AE of special interest (AESI), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wan He, PhD, Principal Investigator — Shenzhen People's Hospital; Keli Zhong, PhD, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China